CLINICAL TRIAL: NCT07204743
Title: Efficacy and Safety of Dapagliflozin in Children With Proteinuria
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Quds University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 382738738
Record Dates: First submitted 2025-09-18; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-08

CONDITIONS: SGLT 2 Inhibitors; Pediatric Kidney Disease; Proteinuric Diseases; Dapagliflozin (Forxiga)
Keywords: Pediatric kidney disease; Safety and efficacy; Kidney function biomarkers; Renal protection; Proteinuria; Dapagliflozin; Pediatric nephrology; SGLT2 inhibitors
MeSH Terms: conditions — Proteinuria | interventions — dapagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dapagliflozin Treatment Arm (Experimental): This arm includes pediatric patients with kidney disease who receive dapagliflozin (5-10 mg daily) as an adjunct therapy. Participants are monitored monthly to assess efficacy and safety outcomes. Key renal function parameters measured include serum creatinine (Cr), blood urea nitrogen (BUN), estimated glomerular filtration rate (eGFR), and 24-hour urinary protein excretion normalized to body surface area. Additional markers such as blood pressure, metabolic status, and potential adverse events (e.g., hypoglycemia, dehydration, urinary tract infections) are also evaluated. The purpose of this arm is to determine the effect of dapagliflozin on reducing proteinuria and improving renal outcomes in the pediatric population.
  Interventions: Drug: Dapagliflozin (5-10 mg daily) - SGLT2 Inhibitor Therapy

INTERVENTIONS:
Drug: Dapagliflozin (5-10 mg daily) - SGLT2 Inhibitor Therapy — Participants will receive dapagliflozin, an oral sodium-glucose cotransporter-2 (SGLT2) inhibitor, administered once daily at a dose of 5-10 mg. The intervention is intended to reduce proteinuria and provide nephroprotection in pediatric patients with kidney disease. Patients will be followed monthly, with monitoring of renal function markers (serum creatinine, blood urea nitrogen, and estimated glomerular filtration rate) and 24-hour urinary protein excretion normalized to body surface area, in addition to safety outcomes such as hypoglycemia, dehydration, and urinary tract infections.

SUMMARY:
This interventional study investigates the efficacy of dapagliflozin, a sodium-glucose co-transporter 2 (SGLT2) inhibitor, in pediatric patients with renal disease. The primary outcomes include changes in 24-hour proteinuria indexed to body surface area (mg/m²/day) and glomerular filtration rate (GFR) before and after dapagliflozin administration. By closely monitoring these parameters, the study aims to assess the renal protective potential of dapagliflozin in children and adolescents.

DETAILED DESCRIPTION:
This is an interventional study designed to evaluate the effect of dapagliflozin, an SGLT2 inhibitor, on renal function in a pediatric population with underlying kidney disease. Eligible participants will include children and adolescents diagnosed with renal impairment.

All participants will receive dapagliflozin at an appropriate pediatric dose and will be followed over the study period. Baseline assessments will include measurement of serum creatinine, blood urea nitrogen (BUN), electrolytes, 24-hour urine protein normalized to body surface area (mg/m²/day), and estimated glomerular filtration rate (eGFR).

Follow-up evaluations will be conducted at regular intervals, with the same laboratory parameters measured to monitor both efficacy and safety. The primary endpoints are:

1. Change in 24-hour proteinuria/m² before and after dapagliflozin therapy.
2. Change in glomerular filtration rate (GFR) before and after treatment.

Secondary endpoints will include trends in serum creatinine, BUN, electrolyte balance, and tolerability of dapagliflozin in this age group. Safety monitoring will be performed throughout the study to detect potential adverse effects, such as hypoglycemia, dehydration, or urinary tract infections.

This study is expected to provide valuable evidence regarding the renal protective effects of dapagliflozin in pediatric patients, contributing to knowledge on its role as a novel therapeutic option in managing pediatric kidney disease.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients aged 4-18 years
* Persistent proteinuria > 500 mg/day despite standard therapy.
* Stable renal function (eGFR ≥ 30 mL/min/1.73 m²).
* Ability to comply with follow-up visits and study procedures.
* Written informed consent obtained from parents or legal guardians, and assent from the patient when appropriate.

Exclusion Criteria:

* Known hypersensitivity or contraindication to dapagliflozin or other SGLT2 inhibitors.
* Severe renal impairment (eGFR < 30 mL/min/1.73 m²) or end-stage renal disease requiring dialysis.
* Active urinary tract infection, severe dehydration, or hypotension.
* Participation in another clinical trial within the last 30 days.
* Any comorbid condition or medical history that, in the investigator's opinion, would interfere with study participation or interpretation of results.

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-08-15 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Comparison of 24-hour proteinuria/m² before and after Dapagliflozin | Baseline to 12 months
Comparison of eGFR before and after Dapagliflozin | Baseline to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Bassil A Leghrouz, MD, Study Director — Al Ahli hospital-Palestine
Locations (1):
- Al Ahli hospital, Hebron, Palestine, Palestinian Territories

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Van Reeth O, Caliment A, de la Fuente Garcia I, Niel O. Safety Profile and Effectiveness of Dapagliflozin in Pediatric Patients with Chronic Kidney Disease. Am J Nephrol. 2024;55(4):463-467. doi: 10.1159/000539300. Epub 2024 May 14. PMID 38735286